CLINICAL TRIAL: NCT06800053
Title: FOCUS ON US: Adapting the FOCUS Program for Sexual and Gender Minority (SGM) Cancer Patients and Caregivers
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was suspended. Lost federal funding due to executive orders.
Sponsor: Charles Kamen (Other)
Collaborators: Wayne State University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Charles Kamen, Ph.D., M.P.H., Assistant professor, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00010099; 1R34CA283408-01 (NIH)
Record Dates: First submitted 2025-01-03; First posted 2025-01-29 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Cancer Support; Oncology Patients; Caregivers
Keywords: Cancer Patients and Caregivers; LGBTQ+

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): This group will complete a baseline assessment and then receive the intervention immediately. Participants will complete a post-intervention assessment survey after completing the intervention. Finally, participants will be contacted for a follow-up assessment 3 months after finishing the intervention.
  Interventions: Behavioral: FOCUS ON US
- Waitlist Control (No Intervention): This group will create a baseline assessment and will not receive the intervention. Participants will complete a post-intervention assessment survey ~3 months after baseline. Following a ~6-month (from baseline) follow-up assessment, this group will be offered the intervention.

INTERVENTIONS:
Behavioral: FOCUS ON US — This intervention will include 5 sessions cover 5 core content areas, represented by the acronym FOCUS. Family involvement (F) Outlook and meaning (O) Coping effectiveness (C) Uncertainty reduction (U) Symptom management (S) Content from every area is presented in the 3 longer in-depth sessions and reinforced in the 2 shorter check-in sessions. FOCUS encourages participants to work as a team, communicate openly, and support one another, and uses skill building (e.g., stress reduction techniques, healthy behaviors), education (e.g., symptom trajectories, information gathering), and problem-solving therapy to address "here-and-now" issues that impact QOL. The intervention is flexible, allowing more attention to be spent on issues relevant to particular patients/caregivers.
  Arms: Intervention

SUMMARY:
Our aim for this study is to assess the feasibility and acceptability and explore potential outcomes of the adapted FOCUS On Us intervention in a two-arm pilot trial. The investigators will randomize 80 sexual and/or gender minority (SGM; e.g., lesbian, gay, bisexual, transgender, queer, etc.) cancer patients and their ≥80 informal caregivers (total N≥160) to either FOCUS On Us (adapted from the evidence-based FOCUS program) or a waitlist control.

ELIGIBILITY:
Inclusion Criteria:

Patients must:

1. have been diagnosed or had a biochemical recurrence or progression of any invasive (e.g., Stage ≥1) cancer within the past 24 months;
2. have at least one informal (unpaid) caregiver willing to participate in the program;
3. identify as a sexual and/or gender minority (SGM) OR have a caregiver who identifies as SGM (e.g., either the patient or caregiver(s) must be SGM);
4. be age 18 or older;
5. be able to complete all written and oral components of the study in English;
6. provide informed consent;
7. live in the United States.

Caregivers must:

1. self-report having provided support for a cancer patient as an informal (unpaid) caregiver;
2. have a cancer patient for whom they provided support willing to participate in the program;
3. identify as a sexual and/or gender minority (SGM) OR have provided support to a patient who identifies as SGM (e.g., either the patient or caregiver(s) must be SGM);
4. be age 18 or older;
5. be able to complete all written and oral components of the study in English;
6. provide informed consent;
7. live in the United States

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | 3 months after randomization
  To assess retention feasibility, we will consider the intervention feasible if ≥75% of participants attend the majority of FOCUS On Us sessions (3 out of 5, 2 of which are longer content sessions), and ≥75% complete post-intervention and 3-month follow-up assessments. The feasibility estimates will be reported as a percentage +/- a 95% confidence interval.
Acceptability | 3 months after randomization
  We will consider the intervention acceptable if 80% of participants are highly satisfied with FOCUS On Us on our satisfaction questionnaire (average rating ≥4 out of a maximum of 5).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Wayne State University, Detroit, Michigan
  - University Of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No